CLINICAL TRIAL: NCT00934973
Title: Management of Irritable Bowel Syndrome in Primary Care: Feasibility Randomised Controlled Trial of Mebeverine, Methylcellulose, Placebo and a Patient Self-management Cognitive Behavioural Therapy Website. (MIBS Trial)
Brief Title: Management of Irritable Bowel Syndrome in Primary Care (MIBS Trial)
Acronym: MIBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hazel Everitt (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Hazel Everitt, Principal Investigator, University of Southampton
Organization: University of Southampton (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 5953; 2009-013426-16 (EudraCT Number)
Record Dates: First submitted 2009-06-29; First posted 2009-07-08 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; treatment
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — mebeverine; Methylcellulose; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- mebeverine + no website (Active Comparator): Mebeverine 135mg tds for 6 weeks
  Interventions: Drug: mebeverine; Behavioral: No website
- methylcellulose + no website (Active Comparator): methylcellulose 3 tablets twice a day for 6 weeks
  Interventions: Drug: methylcellulose; Behavioral: No website
- placebo + no website (Placebo Comparator): placebo tablets
  Interventions: Drug: placebo; Behavioral: No website
- mebeverine + CBT website minimal support (Active Comparator): mebeverine 135mg tds and access to website
  Interventions: Drug: mebeverine; Behavioral: CBT website with minimal support
- methylcellulose + CBT website (Active Comparator): methylellulose 3 tablets twice a day and access to website
  Interventions: Drug: methylcellulose; Behavioral: CBT website with minimal support
- placebo + CBT website minimal support (Placebo Comparator): placebo tablets and access to website
  Interventions: Drug: placebo; Behavioral: CBT website with minimal support
- mebeverine + CBT website with support (Active Comparator): mebeverine 135mg tds and access to website with nurse support session
  Interventions: Drug: mebeverine; Behavioral: CBT website with support
- methylcellulose + CBT website support (Active Comparator): methylcellulose 3 tablets twice a day and access to website with nurse support
  Interventions: Drug: methylcellulose; Behavioral: CBT website with support
- placebo + CBT website with support (Placebo Comparator): placebo tablets and access to website with nurse support
  Interventions: Drug: placebo; Behavioral: CBT website with support

INTERVENTIONS:
Drug: mebeverine — overencapsulated mebeverine 135 mg tds for 6 weeks
  Arms: mebeverine + CBT website minimal support; mebeverine + CBT website with support; mebeverine + no website
Drug: methylcellulose — overencapsulated methylcellulose 3 tablets bd for 6 weeks
  Arms: methylcellulose + CBT website; methylcellulose + CBT website support; methylcellulose + no website
Drug: placebo — overencapsulated placebo tablets 1 tds for 6 weeks
  Arms: placebo + CBT website minimal support; placebo + CBT website with support; placebo + no website
Behavioral: CBT website with support — cognitive behavioral therapy with nurse telephone session and email support
  Arms: mebeverine + CBT website with support; methylcellulose + CBT website support; placebo + CBT website with support
Behavioral: No website — No CBT website
  Arms: mebeverine + no website; methylcellulose + no website; placebo + no website
Behavioral: CBT website with minimal support
  Arms: mebeverine + CBT website minimal support; methylcellulose + CBT website; placebo + CBT website minimal support

SUMMARY:
Aims:

1. To pilot an randomized, controlled trial (RCT) to assess the effectiveness of the commonly prescribed medications in UK general practice for IBS: mebeverine (anti-spasmodic) and methylcellulose (bulking-agent) and of the patient CBT based self-management website.
2. To assess the level of support needed for patients using the patient CBT based self-management website for IBS (i.e., initial 30 minute telephone support session with a nurse and email support or not).

DETAILED DESCRIPTION:
Background:

Irritable bowel syndrome (IBS) affects 10-22% of the United Kingdom (UK) population, with National Health Service (NHS) costs over £200 million a year. Abdominal pain, bloating and altered bowel habit affect quality of life, social functioning and time off work. Current general practitioner (GP) treatment relies on a positive diagnosis, reassurance, lifestyle advice and drug therapies, but many suffer ongoing symptoms.

A recent Cochrane review highlighted the lack of research evidence for IBS drugs. Neither GPs, nor patients have good evidence to inform prescribing decisions. However, IBS drugs are widely used: NHS costs 2005 of nearly £10 million for mebeverine and over £8 million for fiber-based bulking agents.

Cognitive behavioral therapy (CBT) and self-management can be helpful, but poor availability in the NHS restricts its use. Development of web-based CBT could increase access without increased costs.

Plan of Investigation:

135 patients aged 16-60 years with IBS symptoms fulfilling the Rome III criteria, recruited via GP practices, will be randomised to: mebeverine, methylcellulose or placebo for 6 weeks and to the CBT based website with a nurse telephone session and email support, website with minimal support, or no website, thus creating 9 groups.

Outcomes: Irritable bowel symptom severity scale and IBS-QOL will be measured at baseline, 6 and 12 weeks. An intention to treat analysis will be undertaken by analysis of covariance (ANCOVA) for a factorial trial.

Potential Impact:

Development of a web-based self-management CBT program for IBS developed in partnership with patients has the potential to benefit large numbers of patients with low cost to the NHS. CBT has been shown to be of benefit for IBS but it's availability is limited due to the high cost and therapist time required for face-to-face CBT. A website can be accessed at a time and place convenient to the patient and the CBT program undertaken at a pace determined by patient needs. The website could be used as a long term support for self-management.

Determining the effectiveness of commonly used drug treatments will help patients and doctors in making informed treatment decisions regarding the drug management of IBS symptoms, enabling better targeting of treatment to those who may benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 to 60 years with symptoms of irritable bowel syndrome that fulfill the Rome III criteria

Exclusion Criteria:

* Atypical symptoms (unexplained weight loss, rectal bleeding)
* Diagnosis of inflammatory bowel disease, coeliac disease or peptic ulcer disease
* Pregnant or breast feeding
* Currently taking or allergy to mebeverine or methylcellulose

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
IBS Symptom Severity Score | Baseline, 6 and 12 weeks
IBS QOL | Baseline, 6 and 12 weeks
  Quality of life

SECONDARY OUTCOMES:
Subjects Global Assessment of relief | 6 weeks and 12 weeks
  Subjects global assessment of relief
Enablement | 6 and 12 weeks
  Assessment of Enablement
HADs | Baseline, 6 and 12 weeks
  Hospital Anxiety and Depression Score

CONTACTS AND LOCATIONS:
Overall Officials: Hazel A Everitt, MBChB, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Everitt H, Moss-Morris R, Sibelli A, Tapp L, Coleman N, Yardley L, Smith P, Little P. Management of irritable bowel syndrome in primary care: the results of an exploratory randomised controlled trial of mebeverine, methylcellulose, placebo and a self-management website. BMC Gastroenterol. 2013 Apr 21;13:68. doi: 10.1186/1471-230X-13-68. PMID 23602047
- [Result] Everitt HA, Moss-Morris RE, Sibelli A, Tapp L, Coleman NS, Yardley L, Smith PW, Little PS. Management of irritable bowel syndrome in primary care: feasibility randomised controlled trial of mebeverine, methylcellulose, placebo and a patient self-management cognitive behavioural therapy website. (MIBS trial). BMC Gastroenterol. 2010 Nov 18;10:136. doi: 10.1186/1471-230X-10-136. PMID 21087463